CLINICAL TRIAL: NCT00106769
Title: A Phase I Study of the Safety and Immunogenicity of a West Nile Virus Recombinant DNA Plasmid Vaccine, VRC-WNVDNA017-00 VP, in Healthy Adult Volunteers
Brief Title: Vaccine to Prevent West Nile Virus Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 050126; 05-I-0126
Record Dates: First submitted 2005-03-29; First posted 2005-03-30 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-01-15

CONDITIONS: Healthy; West Nile Fever; Healthy Volunteer; HV
Keywords: Flavivirus; Mosquito; Immunity; Preventive; Virus; West Nile Fever; Healthy Volunteer; HV
MeSH Terms: conditions — West Nile Fever; Virus Diseases

INTERVENTIONS:
Drug: VRC-WNVDNA017-00-VP

SUMMARY:
This study will test the safety of an experimental vaccine intended to prevent West Nile virus (WNV) infection and determine if it causes side effects. WNV symptoms may vary from fever and headache, to a polio-like syndrome with paralysis. Infection rarely results in death. The vaccine used in this study contains DNA that instructs the body to produce a small amount of a protein found in WNV. If the body creates resistance or immunity to these proteins, then the vaccine may protect against WNV. Study participants cannot get WNV from the vaccine.

Healthy volunteers between 18 years and 50 years of age may be eligible for this study. Candidates are screened with a medical history, physical examination, and blood and urine tests, including a pregnancy test for women who can become pregnant. Patients undergo the following tests and procedures:

* Vaccine injections: Vaccines are given as injections in the upper arm, using a needleless system called the Biojector 2000. The first injection is on study day 0, the second on day 28 (+/-) 7 days, and the third on day 56 (+/-) 7 days. There must be at least 21 days between injections. The pregnancy test for women of childbearing potential is repeated the day of each vaccine injection.
* Diary card: Participants are given a 5-day diary card after each injection to record their temperature and any symptoms and side effects they may experience for up to 5 days after the injection. The diary cards are returned to the clinic at visits scheduled 2 weeks after each injection. Side effects and symptoms also must be reported immediately to a study nurse or doctor, and a clinic visit may be required for an examination.
* Clinic visits: At day 0 and weeks 2, 4, 6, 8, 10, 12, 24 and 32, participants have a medical history, physical examination (if needed) and blood tests. Vital signs and weight are also recorded. Lymph nodes are examined at day 0 and weeks 2, 4, 6, 8, 10 and 12, and urine samples are collected at day 0 and weeks 2, 4, 6, 8 and 10.

Some of the blood drawn during this study is used for genetic tests to see if different types of immune response to a vaccine are related to genetic differences in people.

DETAILED DESCRIPTION:
Study Design: This is a Phase I open label study to evaluate safety, tolerability, and immune response of a recombinant DNA vaccine, VRC-WNVDNA017-00-VP. The hypothesis is that this regimen will be safe for human administration and elicit immune responses to the West Nile virus. The primary objective is to evaluate the safety and tolerability in humans of the investigational vaccine. Secondary and exploratory objectives are related to the immunogenicity of the study vaccine.

Product Description: VRC-WNVDNA017-00-VP is composed of a single closed circular DNA plasmid that encodes the WNV viral proteins precursor transmembrane (PrM) and envelope (E). Vaccine vials will be supplied at 4 mg/mL. Each DNA vaccination will be 1 mL of vaccine administered intramuscularly (in deltoid muscle) using the Biojector 2000 Needle-Free Injection Management System.

Subjects: Healthy adult volunteers (18 to 50 years old) will be enrolled.

Study Plan: Fifteen volunteers will be enrolled and receive 3 injections on the schedule shown in the schema. The protocol requires nine clinic visits and three telephone follow-up contacts.

Study Duration: 32 weeks clinical follow-up for each participant.

Study Endpoints: The primary endpoint is safety of the regimen; secondary immunogenicity endpoints are an ELISPOT and an intracellular cytokine staining (ICS) assay for WNV-specific T cell responses and a WNV ELISA assay. The principal timepoints for ICS and ELISPOT are Week 0 (baseline), Week 8 and Week 12. ICS and ELISPOT at other study timepoints, as well as other immunogenicity assays through Week 32, will be completed as exploratory evaluations. Stored sera will be tested for WNV neutralizing antibody once an assay is developed.

ELIGIBILITY:
* INCLUSION CRITERIA:

A participant must meet all of the following criteria:

18 to 50 years old.

Available for clinical follow-up through Week 32 of the study.

Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process.

Complete an Assessment of Understanding prior to enrollment and verbalize understanding of all questions answered incorrectly.

Able and willing to complete the informed consent process.

Willing to receive HIV test results and willing to abide by NIH guidelines for partner notification of positive HIV results.

Willing to donate blood for sample storage to be used for future research.

In good general health without clinically significant medical history and has satisfactorily completed screening.

Physical examination and laboratory results without clinically significant findings within the 28 days prior to enrollment.

Laboratory Criteria within 28 days prior to enrollment:

Hemoglobin greater than or equal to 11.5 g/dL for women; greater than or equal to 13.5 g/dL for men.

WBC = 3,300-12,000 cells/mm(3).

Absolute neutrophil count (ANC) within institutional normal range.

Total lymphocyte count greater than or equal to 800 cells/mm(3).

Platelets = 125,000 - 400,000/mm(3).

ALT (SGPT) less than or equal to 1.25 x upper limit of normal.

Serum creatinine less than or equal to 1 x upper limit of normal (less than or equal to 1.3 mg/dL for females; less than or equal to 1.4 mg/dL for males).

Normal urinalysis defined as negative glucose, negative or trace protein, and no clinically significant blood in the urine.

Negative FDA-approved HIV blood test.

Negative Hepatitis B surface antigen.

Negative anti-HCV and negative HCV PCR.

Laboratory Criteria within 12 weeks (84 days) prior to enrollment:

Negative flavivirus serology within 84 days prior to enrollment and no history of prior vaccination against yellow fever or Japanese encephalitis virus.

Female-Specific Criteria:

Negative Beta-HCG pregnancy test (urine or serum) on day of enrollment for women presumed to be of reproductive potential.

A female participant must meet any of the following criteria:

No reproductive potential because of menopause (one year without menses) or because of a hysterectomy, bilateral oophorectomy, or tubal ligation

or

Participant agrees to be heterosexually inactive at least 21 days prior to enrollment and through Week 32 of the study,

or

Participant agrees to consistently practice contraception at least 21 days prior to enrollment and through Week 32 of the study by one of the following methods:

condoms, male or female, with or without a spermicide;

diaphragm or cervical cap with spermicide;

intrauterine device;

contraceptive pills or patch, Norplant, Depo-Provera or other FDA-approved contraceptive method;

male partner has previously undergone a vasectomy for which there is documentation.

EXCLUSION CRITERIA:

A volunteer will be excluded if one or more of the following conditions apply:

Women:

Woman who is breast-feeding or planning to become pregnant during the 32 weeks of study participation.

Volunteer has received any of the following substances:

Immunosuppressive medications or cytotoxic medications or inhaled corticosteroids within the past six months (with the exception of corticosteroid nasal spray for allergic rhinitis or topical corticosteroids for an acute uncomplicated dermatitis);

Blood products within 120 days prior to HIV screening;

Immunoglobulin within 60 days prior to HIV screening;

Investigational research agents within 30 days prior to initial study vaccine administration;

Live attenuated vaccines within 30 days prior to initial study vaccine administration;

Medically indicated subunit or killed vaccines, e.g. influenza, pneumococcal, or allergy treatment with antigen injections, within 14 days of study vaccine administration;

Current anti-TB prophylaxis or therapy.

Volunteer has a history of any of the following clinically significant conditions:

Serious adverse reactions to vaccines such as anaphylaxis, hives, respiratory difficulty, angioedema, or abdominal pain.

Autoimmune disease or immunodeficiency.

Asthma that is unstable or required emergent care, urgent care, hospitalization or intubation during the past two years or that requires the use of oral or intravenous corticosteroids.

Diabetes mellitus (type I or II), with the exception of gestational diabetes.

History of thyroidectomy or thyroid disease that required medication within the past 12 months.

Serious angioedema episodes within the previous 3 years or requiring medication in the previous two years.

Hypertension that is not well controlled by medication or is more than 145/95 at enrollment.

Bleeding disorder diagnosed by a doctor (e.g. factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with IM injections or blood draws.

Malignancy that is active or treated malignancy for which there is not reasonable assurance of sustained cure or malignancy that is likely to recur during the period of the study.

Seizure disorder other than: 1) febrile seizures under the age of two, 2) seizures secondary to alcohol withdrawal more than 3 years ago, or 3) a singular seizure not requiring treatment within the last 3 years.

Asplenia, functional asplenia or any condition resulting in the absence or removal of the spleen.

Allergic reaction to aminoglycoside antibiotics.

Psychiatric condition that precludes compliance with the protocol; past or present psychoses; past or present bipolar disorder; disorder requiring lithium; or within five years prior to enrollment, a history of suicide plan or attempt.

Any medical, psychiatric, social condition, occupational reason or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a volunteer's ability to give informed consent.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15
Dates: Start 2005-03-22; Study Completion 2008-01-15

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Centers for Disease Control and Prevention (CDC). West Nile virus activity--United States, September 29-October 5, 2004. MMWR Morb Mortal Wkly Rep. 2004 Oct 8;53(39):922-3. PMID 15470326
- [Derived] Martin JE, Pierson TC, Hubka S, Rucker S, Gordon IJ, Enama ME, Andrews CA, Xu Q, Davis BS, Nason M, Fay M, Koup RA, Roederer M, Bailer RT, Gomez PL, Mascola JR, Chang GJ, Nabel GJ, Graham BS. A West Nile virus DNA vaccine induces neutralizing antibody in healthy adults during a phase 1 clinical trial. J Infect Dis. 2007 Dec 15;196(12):1732-40. doi: 10.1086/523650. PMID 18190252